CLINICAL TRIAL: NCT00167310
Title: CAD Risk in Schizophrenia: Effect of Omega-3 Fatty Acid Supplementation
Brief Title: Decreasing Risk of Coronary Artery Disease in Schizophrenia by Omega-3 Fatty Acid Supplementation
Acronym: CAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Heart Association (Other); VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Yao, Research Professor of Psychiatry and Pharmaceutical Sciences, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHA 0455676U; VA IRB Protocol ID:02063
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Major Depression; Bipolar Disorder; Coronary Artery Disease
Keywords: Omega-3 fatty acids; Statins; Antipsychotic drug; Antidepressant drug; Antimanic drug; Placebos; Double-blind method; Bipolar (depressed phase)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder; Coronary Artery Disease | interventions — Eicosapentaenoic Acid; Fatty Acids, Omega-3; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Eicosapentaenoic acid (omega-3 fatty acid, 2 g in 4x500 mg softgels daily) + Antipsychotic drug (doctor's choice) treatment for baseline, 1 month, 2 months and 4 months duration.
  Interventions: Drug: Eicosapentaenoic acid (omega-3 fatty acid)
- 2 (Placebo Comparator): Placebo (soy bean oil, 2 g in 4x500 mg softgels daily) + Antipsychotic drug (doctor's choice) treatment for baseline, 1 month, 2 months and 4 months duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eicosapentaenoic acid (omega-3 fatty acid) — 2 g of Eicosapentaenoic acid in 4 x 500 mg capsules daily for baseline, 1 month, 2 months and 4 months
  Other Names: EPA
  Arms: 1
Drug: Placebo — 2 g of Placebo (soy bean oil) in 4 x 500 mg capsules daily for baseline, 1 month, 2 months and 4 months
  Other Names: Soy bean oil
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the administration of omega-3 polyunsaturated fatty acids, particularly eicosapentaenoic acid (EPA), can be useful both to reduce coronary artery disease (CAD) risk and illness severity in clinically-stable patients with schizophrenia (or schizoaffective disorder), major depression or bipolar disorder (depressed phase) being treated with lipid lowering drugs (e.g., statins).

DETAILED DESCRIPTION:
We propose to study the effects of EPA (2 g of EPA in 4 x 500 mg capsules daily) compared to placebo supplementation in clinically-stable schizophrenic patients being treated with statins (n=30 each) for 4 months using a randomized, double-blind design. The National Cholesterol Education Program Adult Treatment Panel III guidelines will be used to select those patients with CAD risk to participate. Clinical assessments and comprehensive assessment of the risk for CAD, including plasma total, high-density lipoprotein (HDL)- (HDL2- and HDL3-), low-density lipoprotein (LDL)- (LDL-Real-, Lp(a)-, and IDL-), and VLDL- (VLDL1,2- and VLDL3-) cholesterol, plasma triglycerides, as well as plasma homocysteine and high sensitivity C-reactive protein, will be conducted at baseline, 1 month, 2 months and 4 months after supplementation. It is anticipated that patients who receive EPA supplementation will have significantly greater reduction in plasma triglycerides and LDL4-cholesterol, and increases in HDL2-cholesterol measures, as well as improvements in psychopathology severity than those patients receiving placebo. If indeed EPA is effective in decreasing the risk of CAD, any psychiatric benefits from EPA supplementation will be a further boon to the patients and the treatment team. A tremendous advantage to the clinical use of EPA includes low cost, no significant side effects, and ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV) criteria for schizophrenia (or schizoaffective disorder), major depression, or bipolar (depressed phase) disorder who are treated with antipsychotic, antidepressant or antimanic drugs and a lipid-lowering drug (statin) for 2 months or longer will be screened to participate in the proposed project.
* Based upon the CAD risk determinants (see below) and the National Cholesterol Education Program (NCEP) recommendation of goals for LDL-lowering therapy, the investigators will only enroll schizophrenic patients with baseline (before statin treatment) LDL-cholesterol exceeding:

  * 70 mg/dL having CAD and CAD risk equivalents, e.g., peripheral arterial disease, abdominal aortic aneurysm, symptomatic carotid artery disease, and diabetes, as well as multiple risk factors that confer a 10-year risk for CAD > 20%
  * 130 mg/dL having 2 or more risk factors; and
  * 160 mg/dL having less than 2 risk factors to participate in the EPA trial.

In addition, these CAD-risk patients have not reached the NCEP goal level within the past year following statin treatment.

* Risk factors for CAD. The NCEP Expert Panel (NIH Publication No. 01-3670, May 2001) on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III or ATPIII) recognizes the following CAD risk factors:

  * being male, 45 years or older, or being female 55 years or older;
  * family history of premature CAD;
  * current cigarette smoking;
  * hypertension with 140/90 mmHg or greater; and
  * low HDL-cholesterol (less than 40 mg/dL).

Exclusion Criteria:

* Patients with history of bleeding disorders, current drug or alcohol abuse (within one month), neurological disorders (including head injury with loss of consciousness for greater than 10 minutes), antisocial personality disorder, borderline personality disorder, or mental retardation as indicated in medical records
* Patients who are pregnant (as determined by urine pregnancy test)
* Patients who have already achieved their NCEP goal in terms of their lipid profile (as indicated in laboratory tests) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K Yao, Ph.D., FACB, Principal Investigator — University of Pittsburgh and VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System (University Drive), Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Fatty Acid: Eicosapentaenoic acid (omega-3 fatty acid, 2 g in 4x500 mg softgels daily) + Antipsychotic drug (doctor's choice) treatment for baseline, 1 month, 2 months and 4 months duration.
  Eicosapentaenoic acid (omega-3 fatty acid): 2 g of Eicosapentaenoic acid in 4 x 500 mg capsules daily for baseline, 1 month, 2 months and 4 months
- Placebo: Placebo (soy bean oil, 2 g in 4x500 mg softgels daily) + Antipsychotic drug (doctor's choice) treatment for baseline, 1 month, 2 months and 4 months duration.
  Placebo: 2 g of Placebo (soy bean oil) in 4 x 500 mg capsules daily for baseline, 1 month, 2 months and 4 months
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid | Placebo
Started | 29 | 28
Completed | 21 | 18
Not Completed | 8 | 10
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Population: The participants withdraw voluntarily after signing the consent form.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acid | Placebo | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8) | 54 (8) | 55 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31 (7) | 31 (6) | 31 (6)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Levels of Triglycerides and Lipoprotein Cholesterol
Description: Biochemical measures: Plasma levels of triglycerides, small dense LDL (LDL3- and LDL4-) cholesterol, large buoyant LDL (LDL1- and LDL2-) cholesterol, and HDL2-cholesterol.
Time Frame: 4 months
Population: Plasma triglyceride levels
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 21 | 18
mg/dL
  Plasma triglyceride | 155 (78) | 182 (67)
  Plasma LDL-1 cholesterol | 12.68 (4.93) | 16.92 (7.10)
  Plasma LDL-2 cholesterol | 14.62 (11.36) | 15.79 (12.37)
  Plasma LDL-3 cholesterol | 40.93 (14.69) | 43.47 (23.44)
  Plasma LDL-4 cholesterol | 15.61 (10.47) | 17.66 (12.50)
  Plasma HDL-2 cholesterol | 8.00 (3.96) | 8.56 (2.41)

2. Secondary Outcome: Plasma Cholesterol Levels in Various Lipoprotein Fractions
Description: Biochemical Measures: Plasma levels of total cholesterol, LDL-cholesterol, HDL-cholesterol, VLDL-cholesterol, Lp(a) cholesterol, IDL-cholesterol, HDL3-cholesterol, VLDL1,2-cholesterol, and VLDL3-cholesterol.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 21 | 18
mg/dL
  Plasma total cholesterol | 158 (38) | 175 (45)
  Plasma LDL cholesterol | 98.14 (30.50) | 109.83 (37.55)
  Plasma HDL cholesterol | 38.95 (11.79) | 40.22 (8.61)
  Plasma VLDL cholesterol | 21.24 (5.27) | 24.67 (6.06)
  Plasma Lp(a) cholesterol | 6.10 (4.06) | 4.83 (2.71)
  Plasma IDL cholesterol | 8.24 (5.70) | 11.17 (6.14)
  Plasma HDL3 cholesterol | 31.00 (8.26) | 31.61 (7.28)
  Plasma VLDL1 + VLDL2 cholesterol | 9.62 (2.85) | 11.45 (3.26)
  Plasma VLDL3 cholesterol | 11.67 (2.82) | 13.39 (3.09)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Omega-3 Fatty Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24
Other Adverse Events (participants affected / at risk) | 2/28 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid (N=28) | Placebo (N=24)
EKG report indicated sinus bradycardia with HR of 39. Patient asymptomatic. (Cardiac disorders) | 1 (1) | 0 (0)
Patient experiences mental problem (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No